CLINICAL TRIAL: NCT00425880
Title: GCRC: Monitoring and Outcome Measures in Asthmatics and Smokers (MOMAS) During Pregnancy
Brief Title: Monitoring and Outcome Measures in Asthmatics and Smokers During Pregnancy
Status: Withdrawn | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0578-F2L; 2K12DA014040-06 (NIH)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Asthma; Tobacco Use
Keywords: Pregnancy; Asthma; Tobacco Abuse; Exhaled Nitric Oxide
MeSH Terms: conditions — Asthma; Tobacco Use; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Pregnant Asthmatics
- Pregnant Smokers
- Healthy Pregnant Controls

SUMMARY:
Asthma and smoking during pregnancy cause significant morbidity in both the mother and the offspring. Asthma represents the most common respiratory disorder during pregnancy and smoking rates during pregnancy range from 15-30% in the United States. Maternal asthma and smoking during pregnancy have been shown to increase the rate of intrauterine growth retardation and preterm delivery, as well as increase the risk of wheeze, asthma, respiratory infections, and otitis media in children. However, controlled asthmatics during pregnancy have similar pregnancy outcomes to non-asthmatic pregnancies. Measurement of the fractional concentration of exhaled nitric oxide (FENO) is a new, easily performed, non-invasive method that has been used to assess airway inflammation in adults and children. The long term goal of this study is to establish baseline FENO values and to monitor airway disease in pregnant asthmatics, pregnant smokers and pregnant controls, and to correlate these levels with other inflammatory markers in the mothers and their offspring. These values will be correlated with current methods to diagnose and monitor disease control in these patients. The use of FENO levels in the pregnant asthmatic may prove to be a better method for monitoring disease control and titrating steroid doses in this population. Finally, this study may identify children at higher risk of developing asthma or allergic disease. This could serve to identify factors that may be modified to prevent or limit the development of these diseases in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be pregnant to participate in the study.
* Patients need to be aged 18 to 35 to participate in the study.
* Smokers must have smoked over 100 cigarettes in their lifetime and currently smoke 5 or more cigarettes per day.
* Asthmatics must be diagnosed with asthma and have a current prescription for an asthma medication such as albuterol or an inhaled steroid.

Exclusion Criteria:

Nonsmokers

* Cannot have smoked more than 100 cigarettes in their lifetime or currently smoke.
* Cannot have any other lung diseases such as asthma, emphysema (COPD), lung cancer, liver disease, cystic fibrosis or other significant respiratory diseases.
* Cannot have been treated with oral steroids or had a respiratory infection in the 4 weeks before study entry.
* Cannot have another illness that can significantly affect quality of life (such as depression or cancer).

Smokers

* Cannot have any other lung diseases such as emphysema (COPD), lung cancer, liver disease, cystic fibrosis or other significant respiratory diseases.
* Cannot have been treated with oral steroids or had a respiratory infection in the 4 weeks before study entry.
* Cannot have another illness that can significantly affect quality of life (such as depression or cancer).

Asthmatics

* Patients in the asthma group cannot have taken theophylline (Theo-24, Theolair, Uniphyl) within 6 months of this study.
* Asthmatics cannot have smoked over 100 cigarettes in their lifetime or be current smokers.
* Cannot have any other lung diseases such as emphysema (COPD), lung cancer, liver disease, cystic fibrosis or other significant respiratory diseases.
* Cannot have been treated with oral steroids or had a respiratory infection in the 4 weeks before study entry.
* Cannot have another illness that can significantly affect quality of life (such as depression or cancer).

All Subjects

* All subjects will be required to avoid antihistamines for 5 days prior to skin testing (can cause false negative results).
* All subjects will be required to avoid food, drink, exercise, and smoking 1 hour prior to exhaled nitric oxide measurement (could falsely increase or decrease levels), and will need to avoid foods that have a high nitrate content for 24 hours prior to exhaled nitric oxide measurement.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from clinics at the University of Kentucky and from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide levels | 9 months

SECONDARY OUTCOMES:
Inhaled corticosteroid dose | 9 months
Asthma control/exacerbations | 9 months
Peripheral blood inflammatory markers | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: James Temprano, M.D., M.H.A., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States